CLINICAL TRIAL: NCT02129296
Title: Intragastric Balloon, Air Versus Fluid Filled: Randomized Prospective Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, PhD, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gastric balloon
Record Dates: First submitted 2014-04-26; First posted 2014-05-02 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Morbid Obesity; Weight Loss; Tolerance
Keywords: Morbid obesity; Gastric balloon; Weight loss; Tolerance; Safety
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hemiosphere® BALLOON (Active Comparator): Balloon filled with air according to the manufacturing company orders 600 or 720 ml air
  Interventions: Device: Air filled balloon
- Fluid filled balloon (Active Comparator): Balloon filled with saline and methylene blue according to the manufacturing company orders
  Interventions: Device: Bioenteric BIB® balloon

INTERVENTIONS:
Device: Air filled balloon — Balloon filled with air according to the manufacturing company orders
  Other Names: first group
  Arms: hemiosphere® BALLOON
Device: Bioenteric BIB® balloon — Balloon filled with saline and methylene blue according to the manufacturing company orders
  Other Names: second group
  Arms: Fluid filled balloon

SUMMARY:
Gastric balloons are an evolving way of reducing weight. There are two types on the market, up to date. Air filled balloons seem to be more safe, and more tolerable.

DETAILED DESCRIPTION:
Morbidly obese patients are categorized into two groups: the 1st group to whom intragastric air filled balloon and the 2nd group to whom saline filled balloon is applied for treatment of their morbid obesity. The aim of study is to compare both types of balloons regarding safety, efficacy and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients

Exclusion Criteria:

* Patient refused
* Non compliant patients
* Psychological patients
* Oesophageal varices, big hiatus hernia, ulcers
* Gastric vascular malformations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Tolerance | 6 months
  Tolerance of the patients toward the balloon regarding vomiting, nausea, dysphagia , gastric pain and dyspepsia

SECONDARY OUTCOMES:
Weight loss | 6 months
  Weight loss by Kg and BMI,
Rate of deflation or puncture | 6 MONTHS
  Rate of deflation or puncture (in air filled, it well be followed up by x ray every 2 weeks while in saline filled, it well be followed up by observation of blue coloured urine

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Abd Ellatif, PhD, Principal Investigator — Mansoura University
Locations (1):
- Hafr Albatin Central hospital, Mansoura University, Egypt